CLINICAL TRIAL: NCT06213883
Title: Characterizing Acute Exercise Response in Restrictive Eating Disorders
Brief Title: Response to Acute Exercise in Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-1585; 1R21MH131787-01A1 (NIH)
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Eating Disorders
Keywords: accelerometer; Adolescent; Aerobic Exercise; Biological Markers; Body Image; Affect; Exercise; Females; Rewards; exercise intensity; restrictive eating
MeSH Terms: conditions — Feeding and Eating Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: Individuals Complete Exercise and Rest Sessions in-lab. We are evaluating the impact of exercise on affect, body image, and biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Response to Exercise and Rest (Experimental): Study participants undergo Prescribed Exercise, Self-Paced Exercise, and Rest conditions over the course of 3 study days
  Interventions: Other: Biobehavioral Response to in-lab exposure to physical activity

INTERVENTIONS:
Other: Biobehavioral Response to in-lab exposure to physical activity — ED severity, biological and affective markers of physical activity response, and both exercise-specific and general positive (reward) and negative (avoidance/escape) valence sensitivities associate with physical activity will be comprehensively examined.

SUMMARY:
Individuals with eating disorders (ED) represent a high-priority clinical population, with among the highest mortality rates of any psychiatric disorder, and driven exercise (DEx) is a symptom evidenced in up to 80% of those with EDs that increases impairment and negatively impacts treatment outcome. This study will develop tasks to characterize cognitive, affective, and biological response to exercise among adolescent and young adult females with EDs and determine whether acute exercise response associates with free-living activity and DEx. This R21 project will provide foundational data to guide research and development of treatments that are more precisely targeted to the symptom of driven exercise and to ultimately improve clinical outcomes associated with EDs.

DETAILED DESCRIPTION:
Eating disorders (EDs) are among the deadliest of all psychiatric disorders. However, first-line treatments for EDs are effective for only roughly 40% of adolescent patients. One barrier to treatment efficacy is the persistence of driven exercise (DEx; exercising in a compulsive manner to control weight and/or regulate emotion), a hallmark symptom reported among many adolescents diagnosed with restrictive EDs (59-73%). Among other negative sequelae, DEx is associated with suicidal behavior, poorer treatment outcome, increased comorbid psychopathology, and risk for relapse. Further, while multiple eating-related tasks have been validated that discriminate between individuals with EDs and healthy populations, there are currently no well-validated tasks that directly assess sensitivity and responsivity to exercise in ED populations. As DEx is a poorly understood symptom that plays a key role in ED maintenance, investigating its biobehavioral underpinnings is of critical importance. Existing research points towards both reward and threat functions of exercise, which may drive and perpetuate DEx among those with EDs. Evaluation of both reward and threat functions of exercise among those with EDs will improve mechanistic understanding of this ED feature; ultimately, improved understanding of DEx will inform treatment targets. The proposed project will recruit adolescent and young adult females (16-25y) with (n = 67) and without (n = 33) EDs from two sites to participate in a comprehensive evaluation of acute exercise response. The current project will 1) characterize variability in biobehavioral response to in-lab exposure to moderate-intensity exercise among those with and without EDs; 2) create and refine tasks that capture engagement of reward- and threat-related systems during exercise; and 3) test hypotheses that acute exercise response is more pronounced among individuals with EDs and that acute exercise response relates to ED symptom severity, DEx, and free-living activity. Detailed explication of acute exercise effects among individuals with EDs in a controlled setting will have significant impact on the empirical study of EDs, specifically to (i) improve assessment of DEx risk and function (ii) elucidate a testable model of DEx risk and (iii) suggest targets for DEx intervention. The methods validated in this project will improve understanding of DEx, a treatment- resistant ED feature. These methods will also lay the groundwork for larger-scale, clinical research which clarifies optimal targets for DEx in ED treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-25
* ED participants must meet full criteria for DSM-5 restrictive-spectrum eating disorders characterized by weight and shape concern, I.e., anorexia nervosa (AN); mild, moderate, or in partial remission), atypical AN, and OSFED -AN type only)
* ED participants must be medically stable, and suitable for outpatient treatment
* Biological Females, Assigned Female at birth
* English Speaking

Exclusion Criteria:

* Those with a medical condition that precludes exercise (e.g., severe asthma) will be excluded for any contraindications

  * Biological Males, Assigned Male at birth
  * BMI less than 16 (over 18 years) or less than 75% expected body weight (under 18 years)
  * Reported intake on Eating Disorder Examination <1000kcal daily
  * Current purging >1x per day
  * Current regular episodes of objective binge eating (>1x/wk)
  * Current self-report of loss-of control eating per the Eating Disorders Examination Interview
  * ED related hospitalization, partial hospitalization, or residential treatment in the past month
  * Any endorsed medical concerns related to physical activity (as probed in the phone screening questions regarding cardiovascular, pulmonary, or metabolic disease).
  * Major medical disorders (e.g., cancer, AIDS)
  * Physical discomfort or difficulty with blood draws
  * Psychotic disorders
  * Intellectual disabilities
  * Developmental disorders
  * Active substance use disorder
  * Current suicidal risk per the Ask Suicide Screening Questionnaire
  * Pregnancy
  * Psychiatric medications that have not been stable for at least 4 weeks
  * Acute sedatives / pain killers (e.g., benzodiazepines, opioids) and prescription stimulants (e.g., methylphenidate, amphetamines) are not permitted for the full day prior to the laboratory session. The noted short-term medication holds only apply to subjects taking the noted medications in cases used to treat ADHD or other psychiatric conditions
  * Resting heart rate <50 beats per minute (assessed at screening visit)
  * Low blood pressure (<90/60), (assessed at screening visit)
  * Daily cannabis use
  * History of light headedness or fainting during blood draws or physical activity
  * History of chest pain during physical activity
  * Bone, joint, cardiac, pulmonary, metabolic, or other medical conditions that may be worsened by physical activity (e.g., COPD, diabetes, hypertension) that are not currently addressed via medication or lifestyle change.
  * Physical disabilities that prohibit task performance (such as blindness or deafness)
  * Any other condition that the investigator believes might put the participant at risk for negative outcomes
  * Individuals with a restrictive eating disorder presentation that does not include weight and shape concern (ARFID) or that has primary binge eating (bulimia nervosa)
  * Indication of health risk associated with exercise on the Physical Activity Readiness Questionnaire

Ages: 16 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Response to in-lab exercise - body image | Every 5 minutes during 30 minute bout of activity . There is no follow up beyond the study day itself.
  the Body Image States Scale is a 6-item scale that asks participants to report on their momentary body satisfaction on a 9-point Likert scale. Each item begins with the sentence "Right now, I feel" [for instance: "Right now, I feel (Extremely dissatisfied to Extremely satisfied) with my physical appearance"]
Response to in-lab exercise - affect | Every 5 minutes during a 30 minute bout of activity. There is no follow up beyond the study day itself.
  Participants self-report items representing the highest loading items from the Physical Activity Affect Scale (PAAS) every 5 minutes during exercise. These items include feeling 'Crummy', 'Enthusiastic', 'Fatigued' and 'Calm'. Participants rate each item using a 5-point scale (0=do not feel-4=feel very strongly).
Response to in-lab exercise - biomarkers | pre-exercise (Baseline), post-exercise (30 minutes), pre-rest (Baseline), post-rest (30 minutes). There is no follow up beyond the study day itself.
  Biomarkers will be collected via blood samples taken before and after exercise and rest and measured via Enzyme-linked immunosorbent assay (ELISA) kits :
  circulating leptin (leptin immunoassay) circulating endocannabinoids (2-arachidonoylglycerol (2-AG) and 2-oleoylglycerol (2-OG) plasma-based immunoassays) circulating brain-derived neurotrophic factor (BDNF immunoassay) circulating cortisol (Cortisol immunoassay)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Project publications will provide full information about procedures and analyses to enable replication. We will share data and code on an institutional webpage for reproducibility.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: At study conclusion

REFERENCES:
- [Background] Schaumberg K, Welch E, Breithaupt L, Hubel C, Baker JH, Munn-Chernoff MA, Yilmaz Z, Ehrlich S, Mustelin L, Ghaderi A, Hardaway AJ, Bulik-Sullivan EC, Hedman AM, Jangmo A, Nilsson IAK, Wiklund C, Yao S, Seidel M, Bulik CM. The Science Behind the Academy for Eating Disorders' Nine Truths About Eating Disorders. Eur Eat Disord Rev. 2017 Nov;25(6):432-450. doi: 10.1002/erv.2553. Epub 2017 Oct 2. PMID 28967161
- [Background] Steinhausen HC. Outcome of eating disorders. Child Adolesc Psychiatr Clin N Am. 2009 Jan;18(1):225-42. doi: 10.1016/j.chc.2008.07.013. PMID 19014869
- [Background] Pisetsky EM, Thornton LM, Lichtenstein P, Pedersen NL, Bulik CM. Suicide attempts in women with eating disorders. J Abnorm Psychol. 2013 Nov;122(4):1042-56. doi: 10.1037/a0034902. PMID 24364606
- [Background] Kolar DR, Gorrell S. A call to experimentally study acute affect-regulation mechanisms specific to driven exercise in eating disorders. Int J Eat Disord. 2020 Dec 1:10.1002/eat.23427. doi: 10.1002/eat.23427. Online ahead of print. PMID 33289120
- [Background] Smith AR, Fink EL, Anestis MD, Ribeiro JD, Gordon KH, Davis H, Keel PK, Bardone-Cone AM, Peterson CB, Klein MH, Crow S, Mitchell JE, Crosby RD, Wonderlich SA, le Grange D, Joiner TE Jr. Exercise caution: over-exercise is associated with suicidality among individuals with disordered eating. Psychiatry Res. 2013 Apr 30;206(2-3):246-55. doi: 10.1016/j.psychres.2012.11.004. Epub 2012 Dec 7. PMID 23219104
- [Background] Dalle Grave R, Calugi S, Marchesini G. Compulsive exercise to control shape or weight in eating disorders: prevalence, associated features, and treatment outcome. Compr Psychiatry. 2008 Jul-Aug;49(4):346-52. doi: 10.1016/j.comppsych.2007.12.007. Epub 2008 Mar 19. PMID 18555054
- [Background] Carter JC, Blackmore E, Sutandar-Pinnock K, Woodside DB. Relapse in anorexia nervosa: a survival analysis. Psychol Med. 2004 May;34(4):671-9. doi: 10.1017/S0033291703001168. PMID 15099421
- [Background] Holtkamp K, Herpertz-Dahlmann B, Hebebrand K, Mika C, Kratzsch J, Hebebrand J. Physical activity and restlessness correlate with leptin levels in patients with adolescent anorexia nervosa. Biol Psychiatry. 2006 Aug 1;60(3):311-3. doi: 10.1016/j.biopsych.2005.11.001. Epub 2005 Dec 27. PMID 16376860
- [Background] Greenwood BN, Foley TE, Le TV, Strong PV, Loughridge AB, Day HE, Fleshner M. Long-term voluntary wheel running is rewarding and produces plasticity in the mesolimbic reward pathway. Behav Brain Res. 2011 Mar 1;217(2):354-62. doi: 10.1016/j.bbr.2010.11.005. Epub 2010 Nov 9. PMID 21070820
- [Background] Sawyer SM, Whitelaw M, Le Grange D, Yeo M, Hughes EK. Physical and Psychological Morbidity in Adolescents With Atypical Anorexia Nervosa. Pediatrics. 2016 Apr;137(4):e20154080. doi: 10.1542/peds.2015-4080. Epub 2016 Mar 29. PMID 27025958
- [Background] Sysko R, Steinglass J, Schebendach J, Mayer LES, Walsh BT. Rigor and reproducibility via laboratory studies of eating behavior: A focused update and conceptual review. Int J Eat Disord. 2018 Jul;51(7):608-616. doi: 10.1002/eat.22900. Epub 2018 Aug 21. PMID 30132949
- [Background] Herring MP, Sailors MH, Bray MS. Genetic factors in exercise adoption, adherence and obesity. Obes Rev. 2014 Jan;15(1):29-39. doi: 10.1111/obr.12089. Epub 2013 Sep 15. PMID 24034448
- [Background] Flack K, Pankey C, Ufholz K, Johnson L, Roemmich JN. Genetic variations in the dopamine reward system influence exercise reinforcement and tolerance for exercise intensity. Behav Brain Res. 2019 Dec 16;375:112148. doi: 10.1016/j.bbr.2019.112148. Epub 2019 Aug 9. PMID 31404557
- [Background] Heyman E, Gamelin FX, Goekint M, Piscitelli F, Roelands B, Leclair E, Di Marzo V, Meeusen R. Intense exercise increases circulating endocannabinoid and BDNF levels in humans--possible implications for reward and depression. Psychoneuroendocrinology. 2012 Jun;37(6):844-51. doi: 10.1016/j.psyneuen.2011.09.017. Epub 2011 Oct 24. PMID 22029953
- [Background] Herring MP, O'Connor PJ, Dishman RK. The effect of exercise training on anxiety symptoms among patients: a systematic review. Arch Intern Med. 2010 Feb 22;170(4):321-31. doi: 10.1001/archinternmed.2009.530. PMID 20177034
- [Background] Greenwood BN, Strong PV, Loughridge AB, Day HE, Clark PJ, Mika A, Hellwinkel JE, Spence KG, Fleshner M. 5-HT2C receptors in the basolateral amygdala and dorsal striatum are a novel target for the anxiolytic and antidepressant effects of exercise. PLoS One. 2012;7(9):e46118. doi: 10.1371/journal.pone.0046118. Epub 2012 Sep 25. PMID 23049953
- [Background] Anderson E, Shivakumar G. Effects of exercise and physical activity on anxiety. Front Psychiatry. 2013 Apr 23;4:27. doi: 10.3389/fpsyt.2013.00027. eCollection 2013. No abstract available. PMID 23630504
- [Background] Asmundson GJ, Fetzner MG, Deboer LB, Powers MB, Otto MW, Smits JA. Let's get physical: a contemporary review of the anxiolytic effects of exercise for anxiety and its disorders. Depress Anxiety. 2013 Apr;30(4):362-73. doi: 10.1002/da.22043. Epub 2013 Jan 8. PMID 23300122
- [Background] Guarda AS, Schreyer CC, Boersma GJ, Tamashiro KL, Moran TH. Anorexia nervosa as a motivated behavior: Relevance of anxiety, stress, fear and learning. Physiol Behav. 2015 Dec 1;152(Pt B):466-72. doi: 10.1016/j.physbeh.2015.04.007. Epub 2015 Apr 3. PMID 25846837
- [Background] Davis C, Kaptein S. Anorexia nervosa with excessive exercise: a phenotype with close links to obsessive-compulsive disorder. Psychiatry Res. 2006 Jun 15;142(2-3):209-17. doi: 10.1016/j.psychres.2005.11.006. Epub 2006 May 12. PMID 16697469
- [Background] Bamber DJ, Cockerill IM, Rodgers S, Carroll D. Diagnostic criteria for exercise dependence in women. Br J Sports Med. 2003;37(5):393-400. doi: 10.1136/bjsm.37.5.393. PMID 14514528
- [Background] Bratland-Sanda S, Martinsen EW, Rosenvinge JH, Ro O, Hoffart A, Sundgot-Borgen J. Exercise dependence score in patients with longstanding eating disorders and controls: the importance of affect regulation and physical activity intensity. Eur Eat Disord Rev. 2011 May-Jun;19(3):249-55. doi: 10.1002/erv.971. PMID 21584917
- [Background] Davis C, Claridge G. The eating disorders as addiction: a psychobiological perspective. Addict Behav. 1998 Jul-Aug;23(4):463-75. doi: 10.1016/s0306-4603(98)00009-4. PMID 9698975
- [Background] Lichtenstein MB, Hinze CJ, Emborg B, Thomsen F, Hemmingsen SD. Compulsive exercise: links, risks and challenges faced. Psychol Res Behav Manag. 2017 Mar 30;10:85-95. doi: 10.2147/PRBM.S113093. eCollection 2017. PMID 28435339
- [Background] Shroff H, Reba L, Thornton LM, Tozzi F, Klump KL, Berrettini WH, Brandt H, Crawford S, Crow S, Fichter MM, Goldman D, Halmi KA, Johnson C, Kaplan AS, Keel P, LaVia M, Mitchell J, Rotondo A, Strober M, Treasure J, Woodside DB, Kaye WH, Bulik CM. Features associated with excessive exercise in women with eating disorders. Int J Eat Disord. 2006 Sep;39(6):454-61. doi: 10.1002/eat.20247. PMID 16637047
- [Background] Davis C, Katzman DK, Kaptein S, Kirsh C, Brewer H, Kalmbach K, Olmsted MP, Woodside DB, Kaplan AS. The prevalence of high-level exercise in the eating disorders: etiological implications. Compr Psychiatry. 1997 Nov-Dec;38(6):321-6. doi: 10.1016/s0010-440x(97)90927-5. PMID 9406737
- [Background] Holtkamp K, Hebebrand J, Herpertz-Dahlmann B. The contribution of anxiety and food restriction on physical activity levels in acute anorexia nervosa. Int J Eat Disord. 2004 Sep;36(2):163-71. doi: 10.1002/eat.20035. PMID 15282686
- [Background] Brewerton TD, Stellefson EJ, Hibbs N, Hodges EL, Cochrane CE. Comparison of eating disorder patients with and without compulsive exercising. Int J Eat Disord. 1995 May;17(4):413-6. doi: 10.1002/1098-108x(199505)17:43.0.co;2-0. PMID 7620482
- [Background] Davis C, Woodside DB. Sensitivity to the rewarding effects of food and exercise in the eating disorders. Compr Psychiatry. 2002 May-Jun;43(3):189-94. doi: 10.1053/comp.2002.32356. PMID 11994836
- [Background] Holtkamp K, Herpertz-Dahlmann B, Mika C, Heer M, Heussen N, Fichter M, Herpertz S, Senf W, Blum WF, Schweiger U, Warnke A, Ballauff A, Remschmidt H, Hebebrand J. Elevated physical activity and low leptin levels co-occur in patients with anorexia nervosa. J Clin Endocrinol Metab. 2003 Nov;88(11):5169-74. doi: 10.1210/jc.2003-030569. PMID 14602745
- [Background] Cook BJ, Wonderlich SA, Mitchell JE, Thompson R, Sherman R, McCallum K. Exercise in Eating Disorders Treatment: Systematic Review and Proposal of Guidelines. Med Sci Sports Exerc. 2016 Jul;48(7):1408-14. doi: 10.1249/MSS.0000000000000912. PMID 26909533
- [Background] Cook B, Leininger L. The ethics of exercise in eating disorders: Can an ethical principles approach guide the next generation of research and clinical practice? J Sport Health Sci. 2017 Sep;6(3):295-298. doi: 10.1016/j.jshs.2017.03.004. Epub 2017 Mar 10. No abstract available. PMID 30356587
- [Background] Hay P, Touyz S, Arcelus J, Pike K, Attia E, Crosby RD, Madden S, Wales J, La Puma M, Heriseanu AI, Young S, Meyer C. A randomized controlled trial of the compuLsive Exercise Activity TheraPy (LEAP): A new approach to compulsive exercise in anorexia nervosa. Int J Eat Disord. 2018 Aug;51(8):999-1004. doi: 10.1002/eat.22920. Epub 2018 Jul 26. PMID 30051623
- [Background] Hausenblas HA, Cook BJ, Chittester NI. Can exercise treat eating disorders? Exerc Sport Sci Rev. 2008 Jan;36(1):43-7. doi: 10.1097/jes.0b013e31815e4040. PMID 18156953
- [Background] Matta Mello Portugal E, Cevada T, Sobral Monteiro-Junior R, Teixeira Guimaraes T, da Cruz Rubini E, Lattari E, Blois C, Camaz Deslandes A. Neuroscience of exercise: from neurobiology mechanisms to mental health. Neuropsychobiology. 2013;68(1):1-14. doi: 10.1159/000350946. Epub 2013 Jun 15. PMID 23774826
- [Background] Dietrich A, McDaniel WF. Endocannabinoids and exercise. Br J Sports Med. 2004 Oct;38(5):536-41. doi: 10.1136/bjsm.2004.011718. PMID 15388533
- [Background] Brellenthin AG, Crombie KM, Hillard CJ, Koltyn KF. Endocannabinoid and Mood Responses to Exercise in Adults with Varying Activity Levels. Med Sci Sports Exerc. 2017 Aug;49(8):1688-1696. doi: 10.1249/MSS.0000000000001276. PMID 28319590
- [Background] Crombie KM, Brellenthin AG, Hillard CJ, Koltyn KF. Psychobiological Responses to Aerobic Exercise in Individuals With Posttraumatic Stress Disorder. J Trauma Stress. 2018 Feb;31(1):134-145. doi: 10.1002/jts.22253. Epub 2018 Feb 1. PMID 29388710
- [Background] Kwan BM, Bryan AD. Affective response to exercise as a component of exercise motivation: Attitudes, norms, self-efficacy, and temporal stability of intentions. Psychol Sport Exerc. 2010 Jan 1;11(1):71-79. doi: 10.1016/j.psychsport.2009.05.010. PMID 20161385
- [Background] Deslandes A, Moraes H, Ferreira C, Veiga H, Silveira H, Mouta R, Pompeu FA, Coutinho ES, Laks J. Exercise and mental health: many reasons to move. Neuropsychobiology. 2009;59(4):191-8. doi: 10.1159/000223730. Epub 2009 Jun 10. PMID 19521110
- [Background] Vankim NA, Nelson TF. Vigorous physical activity, mental health, perceived stress, and socializing among college students. Am J Health Promot. 2013 Sep-Oct;28(1):7-15. doi: 10.4278/ajhp.111101-QUAN-395. Epub 2013 Mar 7. PMID 23470187
- [Background] Chekroud SR, Gueorguieva R, Zheutlin AB, Paulus M, Krumholz HM, Krystal JH, Chekroud AM. Association between physical exercise and mental health in 1.2 million individuals in the USA between 2011 and 2015: a cross-sectional study. Lancet Psychiatry. 2018 Sep;5(9):739-746. doi: 10.1016/S2215-0366(18)30227-X. Epub 2018 Aug 8. PMID 30099000
- [Background] Carek PJ, Laibstain SE, Carek SM. Exercise for the treatment of depression and anxiety. Int J Psychiatry Med. 2011;41(1):15-28. doi: 10.2190/PM.41.1.c. PMID 21495519
- [Background] de Geus EJ, Bartels M, Kaprio J, Lightfoot JT, Thomis M. Genetics of regular exercise and sedentary behaviors. Twin Res Hum Genet. 2014 Aug;17(4):262-71. doi: 10.1017/thg.2014.42. PMID 25034445
- [Background] Klimentidis YC, Raichlen DA, Bea J, Garcia DO, Wineinger NE, Mandarino LJ, Alexander GE, Chen Z, Going SB. Genome-wide association study of habitual physical activity in over 377,000 UK Biobank participants identifies multiple variants including CADM2 and APOE. Int J Obes (Lond). 2018 Jun;42(6):1161-1176. doi: 10.1038/s41366-018-0120-3. Epub 2018 Jun 13. PMID 29899525
- [Background] Watson HJ, Yilmaz Z, Thornton LM, Hubel C, Coleman JRI, Gaspar HA, Bryois J, Hinney A, Leppa VM, Mattheisen M, Medland SE, Ripke S, Yao S, Giusti-Rodriguez P; Anorexia Nervosa Genetics Initiative; Hanscombe KB, Purves KL; Eating Disorders Working Group of the Psychiatric Genomics Consortium; Adan RAH, Alfredsson L, Ando T, Andreassen OA, Baker JH, Berrettini WH, Boehm I, Boni C, Perica VB, Buehren K, Burghardt R, Cassina M, Cichon S, Clementi M, Cone RD, Courtet P, Crow S, Crowley JJ, Danner UN, Davis OSP, de Zwaan M, Dedoussis G, Degortes D, DeSocio JE, Dick DM, Dikeos D, Dina C, Dmitrzak-Weglarz M, Docampo E, Duncan LE, Egberts K, Ehrlich S, Escaramis G, Esko T, Estivill X, Farmer A, Favaro A, Fernandez-Aranda F, Fichter MM, Fischer K, Focker M, Foretova L, Forstner AJ, Forzan M, Franklin CS, Gallinger S, Giegling I, Giuranna J, Gonidakis F, Gorwood P, Mayora MG, Guillaume S, Guo Y, Hakonarson H, Hatzikotoulas K, Hauser J, Hebebrand J, Helder SG, Herms S, Herpertz-Dahlmann B, Herzog W, Huckins LM, Hudson JI, Imgart H, Inoko H, Janout V, Jimenez-Murcia S, Julia A, Kalsi G, Kaminska D, Kaprio J, Karhunen L, Karwautz A, Kas MJH, Kennedy JL, Keski-Rahkonen A, Kiezebrink K, Kim YR, Klareskog L, Klump KL, Knudsen GPS, La Via MC, Le Hellard S, Levitan RD, Li D, Lilenfeld L, Lin BD, Lissowska J, Luykx J, Magistretti PJ, Maj M, Mannik K, Marsal S, Marshall CR, Mattingsdal M, McDevitt S, McGuffin P, Metspalu A, Meulenbelt I, Micali N, Mitchell K, Monteleone AM, Monteleone P, Munn-Chernoff MA, Nacmias B, Navratilova M, Ntalla I, O'Toole JK, Ophoff RA, Padyukov L, Palotie A, Pantel J, Papezova H, Pinto D, Rabionet R, Raevuori A, Ramoz N, Reichborn-Kjennerud T, Ricca V, Ripatti S, Ritschel F, Roberts M, Rotondo A, Rujescu D, Rybakowski F, Santonastaso P, Scherag A, Scherer SW, Schmidt U, Schork NJ, Schosser A, Seitz J, Slachtova L, Slagboom PE, Slof-Op 't Landt MCT, Slopien A, Sorbi S, Swiatkowska B, Szatkiewicz JP, Tachmazidou I, Tenconi E, Tortorella A, Tozzi F, Treasure J, Tsitsika A, Tyszkiewicz-Nwafor M, Tziouvas K, van Elburg AA, van Furth EF, Wagner G, Walton E, Widen E, Zeggini E, Zerwas S, Zipfel S, Bergen AW, Boden JM, Brandt H, Crawford S, Halmi KA, Horwood LJ, Johnson C, Kaplan AS, Kaye WH, Mitchell JE, Olsen CM, Pearson JF, Pedersen NL, Strober M, Werge T, Whiteman DC, Woodside DB, Stuber GD, Gordon S, Grove J, Henders AK, Jureus A, Kirk KM, Larsen JT, Parker R, Petersen L, Jordan J, Kennedy M, Montgomery GW, Wade TD, Birgegard A, Lichtenstein P, Norring C, Landen M, Martin NG, Mortensen PB, Sullivan PF, Breen G, Bulik CM. Genome-wide association study identifies eight risk loci and implicates metabo-psychiatric origins for anorexia nervosa. Nat Genet. 2019 Aug;51(8):1207-1214. doi: 10.1038/s41588-019-0439-2. Epub 2019 Jul 15. PMID 31308545
- [Background] Klein DA, Schebendach JE, Gershkovich M, Bodell LP, Foltin RW, Walsh BT. Behavioral assessment of the reinforcing effect of exercise in women with anorexia nervosa: further paradigm development and data. Int J Eat Disord. 2010 Nov 1;43(7):611-8. doi: 10.1002/eat.20758. PMID 19806608
- [Background] Couturier JL, Lock J. Denial and minimization in adolescents with anorexia nervosa. Int J Eat Disord. 2006 Apr;39(3):212-6. doi: 10.1002/eat.20241. PMID 16485271
- [Background] Solenberger SE. Exercise and eating disorders: a 3-year inpatient hospital record analysis. Eat Behav. 2001 Summer;2(2):151-68. doi: 10.1016/s1471-0153(01)00026-5. PMID 15001043
- [Background] Achamrah N, Coeffier M, Dechelotte P. Physical activity in patients with anorexia nervosa. Nutr Rev. 2016 May;74(5):301-11. doi: 10.1093/nutrit/nuw001. Epub 2016 Apr 6. PMID 27052638
- [Background] Calogero RM, Pedrotty KN. The practice and process of healthy exercise: an investigation of the treatment of exercise abuse in women with eating disorders. Eat Disord. 2004 Winter;12(4):273-91. doi: 10.1080/10640260490521352. PMID 16864521
- [Background] Buhren K, Schwarte R, Fluck F, Timmesfeld N, Krei M, Egberts K, Pfeiffer E, Fleischhaker C, Wewetzer C, Herpertz-Dahlmann B. Comorbid psychiatric disorders in female adolescents with first-onset anorexia nervosa. Eur Eat Disord Rev. 2014 Jan;22(1):39-44. doi: 10.1002/erv.2254. Epub 2013 Sep 12. PMID 24027221
- [Background] Dittmer N, Voderholzer U, Monch C, Cuntz U, Jacobi C, Schlegl S. Efficacy of a Specialized Group Intervention for Compulsive Exercise in Inpatients with Anorexia Nervosa: A Randomized Controlled Trial. Psychother Psychosom. 2020;89(3):161-173. doi: 10.1159/000504583. Epub 2020 Feb 7. PMID 32036375
- [Background] Glashouwer KA, Brockmeyer T, Cardi V, Jansen A, Murray SB, Blechert J, Levinson CA, Schmidt U, Tchanturia K, Wade TD, Svaldi J, Giel KE, Favaro A, Fernandez-Aranda F, Friederich HC, Naumann E, Treasure JL, Tuschen-Caffier B, Vocks S, Werthmann J. Time to make a change: A call for more experimental research on key mechanisms in anorexia nervosa. Eur Eat Disord Rev. 2020 Jul;28(4):361-367. doi: 10.1002/erv.2754. No abstract available. PMID 32567176
- [Background] Meyer C, Taranis L, Goodwin H, Haycraft E. Compulsive exercise and eating disorders. Eur Eat Disord Rev. 2011 May-Jun;19(3):174-89. doi: 10.1002/erv.1122. PMID 21584911
- [Background] Coniglio KA, Cooper M, Selby EA. Behavioral reinforcement of pathological exercise in anorexia nervosa. Int J Eat Disord. 2022 Feb;55(2):184-192. doi: 10.1002/eat.23626. Epub 2021 Oct 9. PMID 34626127
- [Background] Bischoff-Grethe A, McCurdy D, Grenesko-Stevens E, Irvine LE, Wagner A, Yau WY, Fennema-Notestine C, Wierenga CE, Fudge JL, Delgado MR, Kaye WH. Altered brain response to reward and punishment in adolescents with Anorexia nervosa. Psychiatry Res. 2013 Dec 30;214(3):331-40. doi: 10.1016/j.pscychresns.2013.07.004. Epub 2013 Oct 19. PMID 24148909
- [Background] Sala M, Egbert AH, Lavender JM, Goldschmidt AB. Affect, reward, and punishment in anorexia nervosa: a narrative overview. Eat Weight Disord. 2018 Dec;23(6):731-737. doi: 10.1007/s40519-018-0588-9. Epub 2018 Oct 4. PMID 30288725
- [Background] Scharmer C, Gorrell S, Schaumberg K, Anderson D. Compulsive exercise or exercise dependence? Clarifying conceptualizations of exercise in the context of eating disorder pathology. J Clin Sport Psychol. 2020 Jan;46:101586. Epub 2019 Sep 16. PMID 34093941
- [Background] Gorrell S, Schaumberg K, Boswell JF, Hormes JM, Anderson DA. Female Athlete Body Project Intervention with Professional Dancers: A Pilot Trial. Eat Disord. 2021 Jan-Feb;29(1):56-73. doi: 10.1080/10640266.2019.1632592. Epub 2019 Jun 24. PMID 31232675
- [Background] Reilly EE, Dmochowski S, Schaumberg K, Earleywine M, Anderson D. Gender-moderated links between urgency, binge drinking, and excessive exercise. J Am Coll Health. 2016;64(2):104-11. doi: 10.1080/07448481.2015.1085056. PMID 26629729
- [Background] Stiles-Shields C, DclinPsy BB, Lock J, Le Grange D. The effect of driven exercise on treatment outcomes for adolescents with anorexia and bulimia nervosa. Int J Eat Disord. 2015 May;48(4):392-6. doi: 10.1002/eat.22281. Epub 2014 Apr 11. PMID 24729068
- [Background] Stiles-Shields EC, Goldschmidt AB, Boepple L, Glunz C, Le Grange D. Driven exercise among treatment-seeking youth with eating disorders. Eat Behav. 2011 Dec;12(4):328-31. doi: 10.1016/j.eatbeh.2011.09.002. Epub 2011 Sep 16. PMID 22051370
- [Background] Gorrell S, Le Grange D. Update on Treatments for Adolescent Bulimia Nervosa. Child Adolesc Psychiatr Clin N Am. 2019 Oct;28(4):537-547. doi: 10.1016/j.chc.2019.05.002. Epub 2019 Jul 4. PMID 31443872
- [Background] Gorrell S, Loeb KL, Le Grange D. Family-based Treatment of Eating Disorders: A Narrative Review. Psychiatr Clin North Am. 2019 Jun;42(2):193-204. doi: 10.1016/j.psc.2019.01.004. Epub 2019 Apr 3. PMID 31046922
- [Background] Gorrell S, Kinasz K, Hail L, Bruett L, Forsberg S, Lock J, Le Grange D. Rituals and preoccupations associated with bulimia nervosa in adolescents: Does motivation to change matter? Eur Eat Disord Rev. 2019 May;27(3):323-328. doi: 10.1002/erv.2664. Epub 2019 Feb 7. PMID 30734406
- [Background] Gorrell S, Hail L, Kinasz K, Bruett L, Forsberg S, Delucchi K, Lock J, Le Grange D. A test of the DSM-5 severity specifier for bulimia nervosa in adolescents: Can we anticipate clinical treatment outcomes? Int J Eat Disord. 2019 May;52(5):586-590. doi: 10.1002/eat.23034. Epub 2019 Jan 30. PMID 30701572
- [Background] Gorrell S, Matheson BE, Lock J, Le Grange D. Remission in adolescents with bulimia nervosa: Empirical evaluation of current conceptual models. Eur Eat Disord Rev. 2020 Jul;28(4):445-453. doi: 10.1002/erv.2729. Epub 2020 Mar 4. PMID 32130757
- [Background] Schaumberg K, Wonderlich S, Crosby R, Peterson C, Le Grange D, Mitchell JE, Crow S, Joiner T, Bardone-Cone AM. Impulsivity and anxiety-related dimensions in adults with bulimic-spectrum disorders differentially relate to eating disordered behaviors. Eat Behav. 2020 Apr;37:101382. doi: 10.1016/j.eatbeh.2020.101382. Epub 2020 Mar 28. PMID 32247895
- [Background] Schaumberg K, Peters D, Ahrenholtz R, Crombie KM, Zhang R, Gorrell S. Registered report: A pilot investigation of acute exercise response among girls and young women with and without eating disorders. Int J Eat Disord. 2021 Nov;54(11):2057-2065. doi: 10.1002/eat.23587. Epub 2021 Jul 29. PMID 34323294
- [Background] Forbush KT, Wildes JE, Pollack LO, Dunbar D, Luo J, Patterson K, Petruzzi L, Pollpeter M, Miller H, Stone A, Bright A, Watson D. Development and validation of the Eating Pathology Symptoms Inventory (EPSI). Psychol Assess. 2013 Sep;25(3):859-78. doi: 10.1037/a0032639. Epub 2013 Jul 1. PMID 23815116
- [Background] Garner DM, Olmsted MP. Scoring the eating disorder inventory. Am J Psychiatry. 1986 May;143(5):680-1. doi: 10.1176/ajp.143.5.aj1435680. No abstract available. PMID 3457539
- [Background] Meyer C, Plateau CR, Taranis L, Brewin N, Wales J, Arcelus J. The Compulsive Exercise Test: confirmatory factor analysis and links with eating psychopathology among women with clinical eating disorders. J Eat Disord. 2016 Aug 19;4:22. doi: 10.1186/s40337-016-0113-3. eCollection 2016. PMID 27547403
- [Background] Taranis L, Touyz S, Meyer C. Disordered eating and exercise: development and preliminary validation of the compulsive exercise test (CET). Eur Eat Disord Rev. 2011 May-Jun;19(3):256-68. doi: 10.1002/erv.1108. PMID 21584918
- [Background] Horowitz LM, Bridge JA, Teach SJ, Ballard E, Klima J, Rosenstein DL, Wharff EA, Ginnis K, Cannon E, Joshi P, Pao M. Ask Suicide-Screening Questions (ASQ): a brief instrument for the pediatric emergency department. Arch Pediatr Adolesc Med. 2012 Dec;166(12):1170-6. doi: 10.1001/archpediatrics.2012.1276. PMID 23027429
- [Background] Goodman WK, Price LH, Rasmussen SA, Mazure C, Fleischmann RL, Hill CL, Heninger GR, Charney DS. The Yale-Brown Obsessive Compulsive Scale. I. Development, use, and reliability. Arch Gen Psychiatry. 1989 Nov;46(11):1006-11. doi: 10.1001/archpsyc.1989.01810110048007. PMID 2684084
- [Background] Decker JH, Otto AR, Daw ND, Hartley CA. From Creatures of Habit to Goal-Directed Learners: Tracking the Developmental Emergence of Model-Based Reinforcement Learning. Psychol Sci. 2016 Jun;27(6):848-58. doi: 10.1177/0956797616639301. Epub 2016 Apr 15. PMID 27084852
- [Background] Cash TF, Fleming EC, Alindogan J, Steadman L, Whitehead A. Beyond body image as a trait: the development and validation of the Body Image States Scale. Eat Disord. 2002 Summer;10(2):103-13. doi: 10.1080/10640260290081678. PMID 16864251
- [Background] Bohon C, Stice E. Negative affect and neural response to palatable food intake in bulimia nervosa. Appetite. 2012 Jun;58(3):964-70. doi: 10.1016/j.appet.2012.02.051. Epub 2012 Mar 2. PMID 22387716
- [Background] Ellison Z, Foong J, Howard R, Bullmore E, Williams S, Treasure J. Functional anatomy of calorie fear in anorexia nervosa. Lancet. 1998 Oct 10;352(9135):1192. doi: 10.1016/S0140-6736(05)60529-6. No abstract available. PMID 9777839
- [Background] Szuhany KL, Bugatti M, Otto MW. A meta-analytic review of the effects of exercise on brain-derived neurotrophic factor. J Psychiatr Res. 2015 Jan;60:56-64. doi: 10.1016/j.jpsychires.2014.10.003. Epub 2014 Oct 12. PMID 25455510
- [Background] Crombie KM, Cisler JM, Hillard CJ, Koltyn KF. Aerobic exercise reduces anxiety and fear ratings to threat and increases circulating endocannabinoids in women with and without PTSD. Ment Health Phys Act. 2021 Mar;20:100366. doi: 10.1016/j.mhpa.2020.100366. Epub 2020 Nov 2. PMID 34149867
- [Background] Meyer JD, Crombie KM, Cook DB, Hillard CJ, Koltyn KF. Serum Endocannabinoid and Mood Changes after Exercise in Major Depressive Disorder. Med Sci Sports Exerc. 2019 Sep;51(9):1909-1917. doi: 10.1249/MSS.0000000000002006. PMID 30973483
- [Background] Bailer UF, Kaye WH. A review of neuropeptide and neuroendocrine dysregulation in anorexia and bulimia nervosa. Curr Drug Targets CNS Neurol Disord. 2003 Feb;2(1):53-9. doi: 10.2174/1568007033338689. PMID 12769812
- [Background] Klein DA, Mayer LE, Schebendach JE, Walsh BT. Physical activity and cortisol in anorexia nervosa. Psychoneuroendocrinology. 2007 Jun;32(5):539-47. doi: 10.1016/j.psyneuen.2007.03.007. Epub 2007 Apr 25. PMID 17462830
- [Background] Dostalova I, Bartak V, Papezova H, Nedvidkova J. The effect of short-term exercise on plasma leptin levels in patients with anorexia nervosa. Metabolism. 2007 Apr;56(4):497-503. doi: 10.1016/j.metabol.2006.11.008. PMID 17379007
- [Background] Ehrlich S, Salbach-Andrae H, Eckart S, Merle JV, Burghardt R, Pfeiffer E, Franke L, Uebelhack R, Lehmkuhl U, Hellweg R. Serum brain-derived neurotrophic factor and peripheral indicators of the serotonin system in underweight and weight-recovered adolescent girls and women with anorexia nervosa. J Psychiatry Neurosci. 2009 Jul;34(4):323-9. PMID 19568484
- [Background] Ho EV, Klenotich SJ, McMurray MS, Dulawa SC. Activity-Based Anorexia Alters the Expression of BDNF Transcripts in the Mesocorticolimbic Reward Circuit. PLoS One. 2016 Nov 18;11(11):e0166756. doi: 10.1371/journal.pone.0166756. eCollection 2016. PMID 27861553
- [Background] Kumar A, Pareek V, Faiq MA, Ghosh SK, Kumari C. ADULT NEUROGENESIS IN HUMANS: A Review of Basic Concepts, History, Current Research, and Clinical Implications. Innov Clin Neurosci. 2019 May 1;16(5-6):30-37. PMID 31440399
- [Background] Severinsen MCK, Pedersen BK. Muscle-Organ Crosstalk: The Emerging Roles of Myokines. Endocr Rev. 2020 Aug 1;41(4):594-609. doi: 10.1210/endrev/bnaa016. PMID 32393961
- [Background] Schmalbach I, Herhaus B, Passler S, Runst S, Berth H, Wolff-Stephan S, Petrowski K. Cortisol reactivity in patients with anorexia nervosa after stress induction. Transl Psychiatry. 2020 Aug 10;10(1):275. doi: 10.1038/s41398-020-00955-7. PMID 32778654
- [Background] Di Chiara G, Bassareo V, Fenu S, De Luca MA, Spina L, Cadoni C, Acquas E, Carboni E, Valentini V, Lecca D. Dopamine and drug addiction: the nucleus accumbens shell connection. Neuropharmacology. 2004;47 Suppl 1:227-41. doi: 10.1016/j.neuropharm.2004.06.032. PMID 15464140
- [Background] Dubreucq S, Koehl M, Abrous DN, Marsicano G, Chaouloff F. CB1 receptor deficiency decreases wheel-running activity: consequences on emotional behaviours and hippocampal neurogenesis. Exp Neurol. 2010 Jul;224(1):106-13. doi: 10.1016/j.expneurol.2010.01.017. Epub 2010 Feb 4. PMID 20138171
- [Background] Dubreucq S, Durand A, Matias I, Benard G, Richard E, Soria-Gomez E, Glangetas C, Groc L, Wadleigh A, Massa F, Bartsch D, Marsicano G, Georges F, Chaouloff F. Ventral tegmental area cannabinoid type-1 receptors control voluntary exercise performance. Biol Psychiatry. 2013 May 1;73(9):895-903. doi: 10.1016/j.biopsych.2012.10.025. Epub 2012 Dec 11. PMID 23237313
- [Background] Monteleone P, Maj M. Dysfunctions of leptin, ghrelin, BDNF and endocannabinoids in eating disorders: beyond the homeostatic control of food intake. Psychoneuroendocrinology. 2013 Mar;38(3):312-30. doi: 10.1016/j.psyneuen.2012.10.021. Epub 2013 Jan 11. PMID 23313276
- [Background] Leinninger GM, Jo YH, Leshan RL, Louis GW, Yang H, Barrera JG, Wilson H, Opland DM, Faouzi MA, Gong Y, Jones JC, Rhodes CJ, Chua S Jr, Diano S, Horvath TL, Seeley RJ, Becker JB, Munzberg H, Myers MG Jr. Leptin acts via leptin receptor-expressing lateral hypothalamic neurons to modulate the mesolimbic dopamine system and suppress feeding. Cell Metab. 2009 Aug;10(2):89-98. doi: 10.1016/j.cmet.2009.06.011. PMID 19656487
- [Background] Walsh JJ, Tschakovsky ME. Exercise and circulating BDNF: Mechanisms of release and implications for the design of exercise interventions. Appl Physiol Nutr Metab. 2018 Nov;43(11):1095-1104. doi: 10.1139/apnm-2018-0192. Epub 2018 May 18. PMID 29775542
- [Background] Delezie J, Handschin C. Endocrine Crosstalk Between Skeletal Muscle and the Brain. Front Neurol. 2018 Aug 24;9:698. doi: 10.3389/fneur.2018.00698. eCollection 2018. PMID 30197620
- [Background] Hackney AC, Walz EA. Hormonal adaptation and the stress of exercise training: the role of glucocorticoids. Trends Sport Sci. 2013;20(4):165-171. PMID 29882537
- [Background] Willoughby KA, Moore SF, Martin BR, Ellis EF. The biodisposition and metabolism of anandamide in mice. J Pharmacol Exp Ther. 1997 Jul;282(1):243-7. PMID 9223560
- [Background] Fuss J, Steinle J, Bindila L, Auer MK, Kirchherr H, Lutz B, Gass P. A runner's high depends on cannabinoid receptors in mice. Proc Natl Acad Sci U S A. 2015 Oct 20;112(42):13105-8. doi: 10.1073/pnas.1514996112. Epub 2015 Oct 5. PMID 26438875
- [Background] Hagan MM, Havel PJ, Seeley RJ, Woods SC, Ekhator NN, Baker DG, Hill KK, Wortman MD, Miller AH, Gingerich RL, Geracioti TD. Cerebrospinal fluid and plasma leptin measurements: covariability with dopamine and cortisol in fasting humans. J Clin Endocrinol Metab. 1999 Oct;84(10):3579-85. doi: 10.1210/jcem.84.10.6034. PMID 10522999
- [Background] Schwartz MW, Peskind E, Raskind M, Boyko EJ, Porte D Jr. Cerebrospinal fluid leptin levels: relationship to plasma levels and to adiposity in humans. Nat Med. 1996 May;2(5):589-93. doi: 10.1038/nm0596-589. PMID 8616722
- [Background] Zimmer P, Stritt C, Bloch W, Schmidt FP, Hubner ST, Binnebossel S, Schenk A, Oberste M. The effects of different aerobic exercise intensities on serum serotonin concentrations and their association with Stroop task performance: a randomized controlled trial. Eur J Appl Physiol. 2016 Oct;116(10):2025-34. doi: 10.1007/s00421-016-3456-1. Epub 2016 Aug 25. PMID 27562067
- [Background] Kendler KS, Mohs RC, Davis KL. The effects of diet and physical activity on plasma homovanillic acid in normal human subjects. Psychiatry Res. 1983 Mar;8(3):215-23. doi: 10.1016/0165-1781(83)90065-3. PMID 6574541
- [Background] Pizzagalli DA, Evins AE, Schetter EC, Frank MJ, Pajtas PE, Santesso DL, Culhane M. Single dose of a dopamine agonist impairs reinforcement learning in humans: behavioral evidence from a laboratory-based measure of reward responsiveness. Psychopharmacology (Berl). 2008 Feb;196(2):221-32. doi: 10.1007/s00213-007-0957-y. Epub 2007 Oct 2. PMID 17909750
- [Background] Ko IG, Kim CJ, Kim H. Treadmill exercise improves memory by up-regulating dopamine and down-regulating D2 dopamine receptor in traumatic brain injury rats. J Exerc Rehabil. 2019 Aug 28;15(4):504-511. doi: 10.12965/jer.1938316.158. eCollection 2019 Aug. PMID 31523669
- [Background] Eddy MC, Stansfield KJ, Green JT. Voluntary exercise improves performance of a discrimination task through effects on the striatal dopamine system. Learn Mem. 2014 Jun 16;21(7):334-7. doi: 10.1101/lm.034462.114. Print 2014 Jul. PMID 24934332
- [Background] Nagata JM, Carlson JL, Kao JM, Golden NH, Murray SB, Peebles R. Characterization and correlates of exercise among adolescents with anorexia nervosa and bulimia nervosa. Int J Eat Disord. 2017 Dec;50(12):1394-1403. doi: 10.1002/eat.22796. Epub 2017 Nov 7. PMID 29112280
- [Background] Adams R. Revised Physical Activity Readiness Questionnaire. Can Fam Physician. 1999 Apr;45:992, 995, 1004-5. No abstract available. PMID 10216799
- [Background] Lavender JM, De Young KP, Anestis MD, Wonderlich SA, Crosby RD, Engel SG, Mitchell JE, Crow SJ, Peterson CB, Le Grange D. Associations between retrospective versus ecological momentary assessment measures of emotion and eating disorder symptoms in anorexia nervosa. J Psychiatr Res. 2013 Oct;47(10):1514-20. doi: 10.1016/j.jpsychires.2013.06.021. Epub 2013 Jul 20. PMID 23880601
- [Background] Kreidler SM, Muller KE, Grunwald GK, Ringham BM, Coker-Dukowitz ZT, Sakhadeo UR, Baron AE, Glueck DH. GLIMMPSE: Online Power Computation for Linear Models with and without a Baseline Covariate. J Stat Softw. 2013 Sep;54(10):i10. doi: 10.18637/jss.v054.i10. PMID 24403868
- [Background] Dinoff A, Herrmann N, Swardfager W, Lanctot KL. The effect of acute exercise on blood concentrations of brain-derived neurotrophic factor in healthy adults: a meta-analysis. Eur J Neurosci. 2017 Jul;46(1):1635-1646. doi: 10.1111/ejn.13603. Epub 2017 Jun 19. PMID 28493624
- [Background] De Chiara V, Errico F, Musella A, Rossi S, Mataluni G, Sacchetti L, Siracusano A, Castelli M, Cavasinni F, Bernardi G, Usiello A, Centonze D. Voluntary exercise and sucrose consumption enhance cannabinoid CB1 receptor sensitivity in the striatum. Neuropsychopharmacology. 2010 Jan;35(2):374-87. doi: 10.1038/npp.2009.141. PMID 19776732
- [Background] Crombie KM, Sartin-Tarm A, Sellnow K, Ahrenholtz R, Lee S, Matalamaki M, Almassi NE, Hillard CJ, Koltyn KF, Adams TG, Cisler JM. Exercise-induced increases in Anandamide and BDNF during extinction consolidation contribute to reduced threat following reinstatement: Preliminary evidence from a randomized controlled trial. Psychoneuroendocrinology. 2021 Oct;132:105355. doi: 10.1016/j.psyneuen.2021.105355. Epub 2021 Jul 9. PMID 34280820
- [Background] Ehrlich S, Burghardt R, Schneider N, Broecker-Preuss M, Weiss D, Merle JV, Craciun EM, Pfeiffer E, Mann K, Lehmkuhl U, Hebebrand J. The role of leptin and cortisol in hyperactivity in patients with acute and weight-recovered anorexia nervosa. Prog Neuropsychopharmacol Biol Psychiatry. 2009 Jun 15;33(4):658-62. doi: 10.1016/j.pnpbp.2009.03.007. Epub 2009 Mar 16. PMID 19296912
- [Background] Goodwin H, Haycraft E, Meyer C. The relationship between compulsive exercise and emotion regulation in adolescents. Br J Health Psychol. 2012 Nov;17(4):699-710. doi: 10.1111/j.2044-8287.2012.02066.x. Epub 2012 Mar 2. PMID 22385050
- [Background] Allen KL, Byrne SM, Oddy WH, Crosby RD. DSM-IV-TR and DSM-5 eating disorders in adolescents: prevalence, stability, and psychosocial correlates in a population-based sample of male and female adolescents. J Abnorm Psychol. 2013 Aug;122(3):720-32. doi: 10.1037/a0034004. PMID 24016012
- [Background] Lindvall Dahlgren C, Wisting L, Ro O. Feeding and eating disorders in the DSM-5 era: a systematic review of prevalence rates in non-clinical male and female samples. J Eat Disord. 2017 Dec 28;5:56. doi: 10.1186/s40337-017-0186-7. eCollection 2017. PMID 29299311
- [Background] Luking KR, Pagliaccio D, Luby JL, Barch DM. Reward Processing and Risk for Depression Across Development. Trends Cogn Sci. 2016 Jun;20(6):456-468. doi: 10.1016/j.tics.2016.04.002. Epub 2016 Apr 27. PMID 27131776
- [Background] Horowitz LM, Snyder DJ, Boudreaux ED, He JP, Harrington CJ, Cai J, Claassen CA, Salhany JE, Dao T, Chaves JF, Jobes DA, Merikangas KR, Bridge JA, Pao M. Validation of the Ask Suicide-Screening Questions for Adult Medical Inpatients: A Brief Tool for All Ages. Psychosomatics. 2020 Nov-Dec;61(6):713-722. doi: 10.1016/j.psym.2020.04.008. Epub 2020 Apr 28. PMID 32487323
- [Background] Pagliaccio D, Luking KR, Anokhin AP, Gotlib IH, Hayden EP, Olino TM, Peng CZ, Hajcak G, Barch DM. Revising the BIS/BAS Scale to study development: Measurement invariance and normative effects of age and sex from childhood through adulthood. Psychol Assess. 2016 Apr;28(4):429-42. doi: 10.1037/pas0000186. Epub 2015 Aug 24. PMID 26302106
- [Background] Brooks-Gunn J, Warren MP, Rosso J, Gargiulo J. Validity of self-report measures of girls' pubertal status. Child Dev. 1987 Jun;58(3):829-41. PMID 3608653
- [Background] Richson BN, Forbush KT, Chapa DAN, Gould SR, Perko VL, Johnson SN, Christensen KA, Swanson TJ, Tregarthen J. Measurement invariance of the Eating Pathology Symptoms Inventory (EPSI) in adolescents and adults. Eat Behav. 2021 Aug;42:101538. doi: 10.1016/j.eatbeh.2021.101538. Epub 2021 Jul 2. PMID 34247036
- [Background] McCreary DR, Sasse DK. An exploration of the drive for muscularity in adolescent boys and girls. J Am Coll Health. 2000 May;48(6):297-304. doi: 10.1080/07448480009596271. PMID 10863873
- [Background] Dakanalis A, Timko A, Madeddu F, Volpato C, Clerici M, Riva G, Zanetti AM. Are the Male Body Dissatisfaction and Drive for Muscularity Scales reliable and valid instruments? J Health Psychol. 2015 Jan;20(1):48-59. doi: 10.1177/1359105313498108. Epub 2013 Aug 29. PMID 23988678
- [Background] Salbach-Andrae H, Schneider N, Burger A, Pfeiffer E, Lehmkuhl U, Holzhausen M. [Psychometric properties of the Eating Disorder Inventory (EDI-2) in adolescents]. Z Kinder Jugendpsychiatr Psychother. 2010 May;38(3):219-28. doi: 10.1024/1422-4917/a000035. German. PMID 20464663
- [Background] Clausen L, Rosenvinge JH, Friborg O, Rokkedal K. Validating the Eating Disorder Inventory-3 (EDI-3): A Comparison Between 561 Female Eating Disorders Patients and 878 Females from the General Population. J Psychopathol Behav Assess. 2011 Mar;33(1):101-110. doi: 10.1007/s10862-010-9207-4. Epub 2010 Oct 19. PMID 21472023
- [Background] Baker JH, Brosof LC, Munn-Chernoff MA, Lichtenstein P, Larsson H, Maes HH, Kendler KS. Associations Between Alcohol Involvement and Drive for Thinness and Body Dissatisfaction in Adolescent Twins: A Bivariate Twin Study. Alcohol Clin Exp Res. 2018 Nov;42(11):2214-2223. doi: 10.1111/acer.13868. Epub 2018 Sep 4. PMID 30252141
- [Background] Kelley CC, Neufeld JM, Musher-Eizenman DR. Drive for thinness and drive for muscularity: opposite ends of the continuum or separate constructs? Body Image. 2010 Jan;7(1):74-7. doi: 10.1016/j.bodyim.2009.09.008. Epub 2009 Nov 26. PMID 19944659
- [Background] Goodwin H, Haycraft E, Taranis L, Meyer C. Psychometric evaluation of the compulsive exercise test (CET) in an adolescent population: links with eating psychopathology. Eur Eat Disord Rev. 2011 May-Jun;19(3):269-79. doi: 10.1002/erv.1109. PMID 21584919
- [Background] Young S, Touyz S, Meyer C, Arcelus J, Rhodes P, Madden S, Pike K, Attia E, Crosby RD, Wales J, Hay P. Validity of Exercise Measures in Adults with Anorexia Nervosa: The EDE, Compulsive Exercise Test and Other Self-Report Scales. Int J Eat Disord. 2017 May;50(5):533-541. doi: 10.1002/eat.22633. Epub 2016 Oct 3. PMID 27696468
- [Background] Muris P, Merckelbach H, Ollendick T, King N, Bogie N. Three traditional and three new childhood anxiety questionnaires: their reliability and validity in a normal adolescent sample. Behav Res Ther. 2002 Jul;40(7):753-72. doi: 10.1016/s0005-7967(01)00056-0. PMID 12074371
- [Background] Scahill L, Riddle MA, McSwiggin-Hardin M, Ort SI, King RA, Goodman WK, Cicchetti D, Leckman JF. Children's Yale-Brown Obsessive Compulsive Scale: reliability and validity. J Am Acad Child Adolesc Psychiatry. 1997 Jun;36(6):844-52. doi: 10.1097/00004583-199706000-00023. PMID 9183141
- [Background] Goodman WK, Price LH, Rasmussen SA, Mazure C, Delgado P, Heninger GR, Charney DS. The Yale-Brown Obsessive Compulsive Scale. II. Validity. Arch Gen Psychiatry. 1989 Nov;46(11):1012-6. doi: 10.1001/archpsyc.1989.01810110054008. PMID 2510699
- [Background] Berg KC, Peterson CB, Frazier P, Crow SJ. Psychometric evaluation of the eating disorder examination and eating disorder examination-questionnaire: a systematic review of the literature. Int J Eat Disord. 2012 Apr;45(3):428-38. doi: 10.1002/eat.20931. Epub 2011 Jul 8. PMID 21744375
- [Background] Binford RB, Le Grange D, Jellar CC. Eating Disorders Examination versus Eating Disorders Examination-Questionnaire in adolescents with full and partial-syndrome bulimia nervosa and anorexia nervosa. Int J Eat Disord. 2005 Jan;37(1):44-9. doi: 10.1002/eat.20062. PMID 15690465
- [Background] Wade TD, Byrne S, Bryant-Waugh R. The eating disorder examination: norms and construct validity with young and middle adolescent girls. Int J Eat Disord. 2008 Sep;41(6):551-8. doi: 10.1002/eat.20526. PMID 18433026
- [Background] Byrne SM, Allen KL, Lampard AM, Dove ER, Fursland A. The factor structure of the eating disorder examination in clinical and community samples. Int J Eat Disord. 2010 Apr;43(3):260-5. doi: 10.1002/eat.20681. PMID 19350647
- [Background] Sullivan-Toole H, DePasque S, Holt-Gosselin B, Galvan A. Worth working for: The influence of effort costs on teens' choices during a novel decision making game. Dev Cogn Neurosci. 2019 Jun;37:100652. doi: 10.1016/j.dcn.2019.100652. Epub 2019 Apr 30. PMID 31075712
- [Background] Cook B, Hausenblas H, Freimuth M. Exercise addiction and compulsive exercising: Relationship to eating disorders, substance use disorders, and addictive disorders. In: Eating Disorders, Addictions, and Substance Use Disorders. Eating Disorders. ; 2014:127-144.
- [Background] Adams J. Understanding exercise dependence. J Contemp Psychother. 2009;39:231-240.
- [Background] Adams J, Kirkby RJ. Excessive exercise as an addiction: A review. Addict Res Theory. Published online 2002.
- [Background] Fortier MS, Sweet SN, O'Sullivan TL, Williams GC. A self-determination process model of physical activity adoption in the context of a randomized controlled trial. Psychol Sport Exerc. 2007;8(5):741-757.
- [Background] Zerwas S, Yilmaz Z, Crowley J, et al. Anorexia nervosa and obsessive compulsive disorder polygenic risk score: Associations with adolescent eating disorder phenotypes. Pap Present World Congr Psychiatr Genet. Published online 2017.
- [Background] Le Grange D, Eisler I. The link between anorexia nervosa and excessive exercise: A review. Eur Eat Disord Rev. 1993;1(2):100-119. doi:10.1002/erv.2400010205
- [Background] Cooper Z, Fairburn C. Eating Disorder Examination. Published online September 12, 2011. doi:10.1037/t03975-000
- [Background] McCreary DR, Sasse DK, Saucier DM, Dorsch KD. Measuring the Drive for Muscularity: Factorial Validity of the Drive for Muscularity Scale in Men and Women. Psychol Men Masculinity. 2004;5(1):49-58. doi:10.1037/1524-9220.5.1.49
- [Background] Beck AT, Steer RA, Brown G. Beck Depression Inventory-II. Published online September 12, 2011. doi:10.1037/t00742-000
- [Background] Spielberger CD. State-Trait Anxiety Inventory. In: Weiner IB, Craighead WE, eds. The Corsini Encyclopedia of Psychology. John Wiley & Sons, Inc.; 2010:corpsy0943. doi:10.1002/9780470479216.corpsy0943
- [Background] Cooper A, Gomez R. The Development of a Short Form of the Sensitivity to Punishment and Sensitivity to Reward Questionnaire. J Individ Differ. 2008;29(2):90-104. doi:10.1027/1614-0001.29.2.90
- [Background] Carver CS, White TL. Behavioral inhibition, behavioral activation, and affective responses to impending reward and punishment: The BIS/BAS Scales. J Pers Soc Psychol. 1994;67:319-333. doi:10.1037/0022-3514.67.2.319
- [Background] Torrubia R, Tobeña A. A scale for the assessment of "susceptibility to punishment" as a measure of anxiety: Preliminary results. Personal Individ Differ. 1984;5:371-375. doi:10.1016/0191-8869(84)90078-3
- [Background] Torrubia R, Ávila C, Moltó J, Caseras X. The Sensitivity to Punishment and Sensitivity to Reward Questionnaire (SPSRQ) as a measure of Gray's anxiety and impulsivity dimensions. Personal Individ Differ. 2001;31(6):837-862. doi:10.1016/S0191-8869(00)00183-5
- [Background] Tiggemann M, Miller J. The Internet and Adolescent Girls' Weight Satisfaction and Drive for Thinness. Sex Roles. 2010;63(1):79-90. doi:10.1007/s11199-010-9789-z
- [Background] Balsamo M, Romanelli R, Innamorati M, Ciccarese G, Carlucci L, Saggino A. The State-Trait Anxiety Inventory: Shadows and Lights on its Construct Validity. J Psychopathol Behav Assess. 2013;35(4):475-486. doi:10.1007/s10862-013-9354-5